CLINICAL TRIAL: NCT03375710
Title: A Prospective, Multi-Center, Open-Label, Single-Arm Clinical Trial Evaluating the Safety and Efficacy of the Cordella™ Heart Failure System in (New York Heart Association) NYHA Class III Heart Failure Patients
Brief Title: SIRONA Trial Heart Failure NYHA Class III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endotronix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ETX-HFS-PA-01
Record Dates: First submitted 2017-12-07; First posted 2017-12-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure NYHA Class III
Keywords: Heart Failure; Heart Diseases; Cardiovascular Disease
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cordella™ Heart Failure System (Experimental): Cordella™ Heart Failure System and implant of Cordella™ Pulmonary Artery Sensor System (CorPASS)
  Interventions: Device: Cordella™ Heart Failure System

INTERVENTIONS:
Device: Cordella™ Heart Failure System — The Cordella™ Heart Failure System collects, records, and transmits physiologic data and communications from the patient at home to clinicians for assessment, patient communication, and patient-centered heart failure management. The system consists of the following components:
  1. myCordella™ Patient Management Portal
  2. myCordella™ Hub
  3. myCordella™ Peripherals, including the Cordella™ Pulmonary Artery Sensor System (CorPASS)

SUMMARY:
This is a prospective, multi-center, open-label, single-arm feasibility trial to assess device safety and efficacy of the Cordella™ Heart Failure System in 10 NYHA Class III heart failure patients who will receive the Cordella™ Sensor implant.

DETAILED DESCRIPTION:
The objectives of this study are to establish that the Cordella™ Sensor can be safely delivered, deployed, and remain stable within the target pulmonary artery (PA) segment through 30 days post-implant as well as to measure the accuracy of Cordella™ Sensor PA pressure measurements compared with fluid-filled catheter PA pressure measurements obtained by standard right heart catheterization (RHC) at 90 days post implant. Safety measures will include the frequency and rates of adverse events, both overall and for each specific event, which will be collected throughout the study. Subjects will remain in this trial for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent
2. Male or female, at least 18 years of age
3. Diagnosis of HF ≥ 3 months with either preserved or reduced left ventricular ejection fraction (LVEF)
4. Diagnosis of NYHA Class III HF at the time of Screening with at least 1 HF-related hospitalization, HF treatment in a hospital day-care setting, or urgent outpatient clinic HF visit within the last year
5. Subjects must be receiving appropriate medical management of HF for 3 months prior to Screening and clinically stable for at least 1 month prior to study entry
6. Subjects with a Body Mass Index (BMI) < 35 kg/mL2 and chest circumference < 1050 mm
7. Subjects with right pulmonary artery branch diameter sized between 14 mm and 20 mm (target Sensor implant site) over a length of at least 30mm
8. Subjects with distance between target implant site (right PA branch) and ventral thoracic skin surface of < 12cm
9. Subjects who are physically able to hold the myCordella™ Patient Reader unit (approximate weight 600g) against the ventral thoracic surface for up to 2 minutes per day while in a seated. position, as well as dock and undock the myCordella™ Patient Reader
10. Subjects with sufficient eyesight, hearing, and mental capacity to respond to the myCordella™ Patient Reader's audio/visual cues and operate the myCordella™ Patient Reader.
11. Subject has sufficient Cellular and/ or Wi- Fi Internet coverage at home
12. Subject agrees to return to the treating Investigator for all scheduled follow up visits and can return to the hospital for follow up
13. Subject compliance as defined by data collection and transmissions at least 5 days a week (does not have to be consecutive days) using the myCordella™ Hub & Peripherals for at least 1 week during the screening period

Exclusion Criteria:

1. Subjects with primary pulmonary hypertension.
2. Subjects with an active infection at the Sensor Implant Visit
3. Subjects with history of recurrent (> 1) pulmonary embolism or deep vein thrombosis
4. Subjects who have had a major cardiovascular event (e.g., myocardial infarction, stroke) within 2 months of the Screening Visit
5. Subjects whereby RHC or computed tomography pulmonary angiography (CTPA) is contraindicated
6. Subjects with a Cardiac Resynchronization Device (CRT), Internal Cardiac Defibrillator (ICD) or pacemaker (if implanted less than 6 months or has more than a single lead), or Left Ventricular Assist Device (LVAD)
7. Any major surgery within 30 days of the Sensor Implant Visit.
8. Subjects with a Glomerular Filtration Rate (GFR) <30 ml/min or who are on chronic renal dialysis
9. Specific liver enzymes [Aspartate Aminotransferase (AST) (SGOT), and Alanine Aminotransferase (ALT) (SGPT) >3 times the upper limit of normal
10. Subjects likely to undergo lung and/ or heart transplantation within 24 months of the Screening Visit.
11. Subjects with congenital heart disease or mechanical/tissue right heart valve(s)
12. Subjects with known coagulation disorders
13. Subjects with a hypersensitivity or allergy to platelet aggregation inhibitors including aspirin, clopidogrel, prasugrel, and ticagrelor; or patients unable to take dual antiplatelet or anticoagulants for one month post implant
14. Subjects enrolled in another investigational trial.
15. Known history of life threatening allergy to contrast dye.
16. Subjects who are unwilling or deemed by the Investigator to be unwilling to comply with the study protocol, or subjects with a history of non-compliance
17. Subjects with large metal implants/prostheses or any other materials in the thoracic cavity that may interfere with the Cordella™ Pulmonary Artery Sensor System performance
18. Subjects with an indwelling inferior vena cava (IVC) filter
19. Subjects who are pregnant or breastfeeding
20. Subjects whose clinical condition, in the opinion of the Investigator, makes them an unsuitable candidate for the study
21. Severe illness, other than heart disease, which would limit survival to <1 year
22. Subjects who have had intractable arrhythmias within 2 month of the Screening Visit
23. Subjects with patent foramen ovale (PFO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Safety Freedom form Adverse events | 30 days
  Freedom from adverse events associated with use of the Cordella™ HF System
Efficacy: Accuracy | 90 days
  Accuracy of Cordella™ Sensor PA pressure measurements, compared to standard-of-care fluid-filled catheter PA pressure measurements obtained by standard Right Heart Catheter

SECONDARY OUTCOMES:
Frequency of Adverse Events | 30 days and 2 years
  Frequency of adverse events throughout the study
Device/system-related complications | 30 days and 2 years
  Device/system-related complications
Pressure sensor failure rate | 30 days and 2 years
  Pressure sensor failure rate throughout the study
Accuracy of Cordella™ sensor pressure measurements | 2 years
  Accuracy of Cordella™ Sensor PA pressure measurements compared with echo pulmonary artery pressure (PAP) measurements
Percentage of device success | 90 days
  Percentage of device success as documented by ability of the System to successfully transmit collected data to a secure database
Change in Pulmonary Artery (PA) pressure | 90 days
  Change in PA pressure pre- and post-implant
Heart Failure (HF) Hospitalizations | 90 days
  Frequency of HF hospitalizations, HF treatments in a hospital day-care setting, or urgent outpatient clinic HF visits.
Quality of Life measured by Kansas City Cardiomyopathy Questionnaire | 90 days and 2 years
  Quality of Life measured by KCCQ at 90 days and 2 years post implant procedure
Quality of Life measured by EuroQOL EQ-5D-5L | 90 days and 2 years
  Quality of Life measured by EuroQOL EQ-5D-5L at 90 days and 2 years post implant procedure
Adherence to regular myCordella™ Peripherals measurements | 90 days and 2 years
  Adherence to regular myCordella™ Peripherals measurements

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sauerland, Study Director — Endotronix, Inc.
Locations (2):
- Ziekenhuis Oost Limburg, Genk, Belgium
- Galway University Hospital, Galway, Ireland